CLINICAL TRIAL: NCT04893122
Title: Impact of the COVID-19 Pandemic on Emergency Department Attendances and Admissions in Southampton for Children and Young Adults
Brief Title: Impact of Pandemic of Presentation to Emergency Department and Admissions
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 63328
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Emergencies
Keywords: emergencies; children; adolescents; young adult
MeSH Terms: conditions — Emergencies | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 pandemic — Study focuses on the impact of the COVID-19 pandemic on emergency attendances and admissions.

SUMMARY:
Observational study assessing the impact of the COVID-19 pandemic on presentations and admission to hospital in children and young adults.

DETAILED DESCRIPTION:
The COVID-19 pandemic has had a major impact on healthcare utilisation and delivery for children and young adults. This is despite these groups experiencing minimal morbidity and almost no mortality as a direct result of the pandemic. The immediate impact of the first lockdown in April 2020 has been well documented. A number of studies show a marked reduction in presentations of children and young adults to the emergency department.

The question is now, are these trends continuing and are they particularly impacting on specific groups and on specific presentations? With these data, services can be modified to minimise any potential for deleterious effects. It may also be possible to target groups who are not utilising health services as the investigators would expect.

The investigators will use fully anonymised routine data on presentations and admission of 0 to 24 years olds to University Hospital Southampton NHS Foundation Trust. Data will be graphed to show trends in activity before and after the start of the pandemic. An interrupted time series regression analysis will be used to assess the significance of any changes in trends.

ELIGIBILITY:
Inclusion Criteria:

* Children and young adults aged 0 to 24 years
* Presented +/- admitted to the emergency department at University Hospital Southampton NHS Foundation Trust between the 1st of April 2016 and 31st of March 2021

Exclusion Criteria: None

Ages: 0 Years to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and young adults aged 0 to 24 years who have presented +/- admitted to the emergency department at University Hospital Southampton NHS Foundation Trust between the 1st of April 2016 and 31st of March 2021. Some children presented to paediatric assessment unit prior to September 2019; after that the patient pathway was merged with the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 166459 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Attendance in emergency department or paediatric assessment unit | 5 years from April 2016
  Attendance at the emergency department in Southampton defined as being booked onto the emergency department admission system.

SECONDARY OUTCOMES:
Emergency admission to hospital | 5 years from April 2016
  Admission to University Hospital Southampton NHS Foundation Trust defined as being in hospital for more than four hours. Participants will be divided into the same subgroups as per attendances.

IPD SHARING:
Plan to Share IPD: No
No ethics approval.

REFERENCES:
- [Derived] Solanke F, Easton S, Selby A, James D, Roberts G. Impact of COVID-19 pandemic on emergency department attendances for young people. Arch Dis Child. 2023 May 3;107(10):e1-e7. doi: 10.1136/archdischild-2021-323389. PMID 35551049

DOCUMENTS (1):
  • Study Protocol (2021-02-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT04893122/Prot_000.pdf